CLINICAL TRIAL: NCT04619407
Title: Screening for SARS-CoV-2-Infections in Teachers, Childcare Educators, Pupils and Preschoolers in the State of Mecklenburg-Vorpommern
Brief Title: Screening for COVID-19 in Teachers, Childcare Educators, Pupils and Preschoolers
Acronym: COKITS
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: Ministry of Education, Science and Culture of the State of Mecklenburg-Vorpommern (Unknown); Ministry of Social Affairs, Integration and Equality of the State of Mecklenburg-Vorpommern (Unknown); State Office for Health and Social Affairs of the State of Mecklenburg-Vorpommern (Unknown)
Responsible Party: Sponsor
Other Study IDs: BB 179/20
Record Dates: First submitted 2020-11-04; First posted 2020-11-06 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV-2
Keywords: serology; antibody formation; epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, nasal/throat swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- teacher: * Employed in a school in Mecklenburg-Vorpommern
  * Age between 18 to 67 years
  * Willing and able to provide informed consent
  * Over 5 months: Monthly nasopharyngeal swabs for SARS-CoV-2 PCR, additionally blood samples for SARS-CoV-2 antibody testing will be taken at the beginning and at the end of the study
  Interventions: Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Serum testing
- pupils: * Attending school in Mecklenburg-Vorpommern
  * Age between 6 to 17 years
  * Agreement to participate
  * Legal representative willing and able to provide informed consent
  * Over 5 months: Monthly nasopharyngeal swabs for SARS-CoV-2 PCR
  Interventions: Diagnostic Test: Nasopharyngeal swab
- childcare educators: * Employed in a kindergarten in Mecklenburg-Vorpommern
  * Age between 18 to 67 years
  * Willing and able to provide informed consent
  * Over 5 months: Monthly nasopharyngeal swabs for SARS-CoV-2 PCR, additionally blood samples for SARS-CoV-2 antibody testing will be taken at the beginning and at the end of the study
  Interventions: Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Serum testing
- preschoolers: * Attending kindergarten in Mecklenburg-Vorpommern
  * Age between 3 to 6 years
  * Agreement to participate
  * Legal representative willing and able to provide informed consent
  * Over 5 months: Monthly nasopharyngeal swabs for SARS-CoV-2 PCR
  Interventions: Diagnostic Test: Nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab — SARS-CoV-2 PCR
Diagnostic Test: Serum testing — Anti-SARS-CoV-2 antibody testing (IgA and IgG ELISA)
  Groups: childcare educators; teacher

SUMMARY:
The main objectives of this study are

1. to establish the prevalence of SARS-CoV-2 in schools and kindergartens in the State of Mecklenburg-Vorpommern in autumn and winter 2020/2021
2. to monitor the future spread of the disease by assessing serological responses to SARS-CoV-2 in teachers and childcare educators over time

DETAILED DESCRIPTION:
Detailed Description:

This study aims to collect information on teachers and childcare educators as well as on pupils and preschoolers in the State of Mecklenburg-Vorpommern

Over a 5 month period, 5 study visits per participant are planned. At each visit, nasal/throat swabs (for PCR testing) will be collected and participants will be asked to fill in a questionnaire (asking for SARS-CoV-2 risk factors, perceived risk, and impact of the pandemic on their quality of life). In adults, additional blood samples (for SARS-CoV-2 antibody testing) will be collected at the first and the last study visit. This will help to gain a better understanding of viral load and antibody development over time.

The remaining blood samples will be stored in a repository for future research.

The study is part of a modular SARS-CoV-2-research programme of the University Medicine Greifswald.

ELIGIBILITY:
Inclusion criteria:

* See cohort descriptions
* Willing to have blood samples stored for future research

Exclusion criteria:

- None

Ages: 3 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Teachers and childcare educators as well as pupils and preschoolers
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Share of participants with SARS-CoV-2 detectable in PCR | 5 months
  Percentage of SARS-CoV-2 PCR positive participants (children and educational staff)

SECONDARY OUTCOMES:
Seroprevalence of SARS-CoV-2 antibodies | At study inclusion
  Percentage of Anti-SARS-COV2 S protein IgA and IgA ELISA positive participants (educational staff)
Seroprevalence of SARS-CoV-2 antibodies | 5 months
  Percentage of Anti-SARS-COV2 S protein IgA and IgA ELISA positive participants (educational staff)
SARS-CoV-2 risk factors, perceived risk of infection, and impact of the pandemic on quality of life | At study inclusion
  As assessed by a monthly questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, and impact of the pandemic on quality of life | 1 month
  As assessed by a monthly questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, and impact of the pandemic on quality of life | 2 months
  As assessed by a monthly questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, and impact of the pandemic on quality of life | 3 months
  As assessed by a monthly questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, and impact of the pandemic on quality of life | 4 months
  As assessed by a monthly questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, and impact of the pandemic on quality of life | 5 months
  As assessed by a monthly questionnaire
Share of participants with SARS-CoV-2 detectable in PCR | At study inclusion
  Percentage of SARS-CoV-2 PCR positive participants (children and educational staff)
Share of participants with SARS-CoV-2 detectable in PCR | 1 month
  Percentage of SARS-CoV-2 PCR positive participants (children and educational staff)
Share of participants with SARS-CoV-2 detectable in PCR | 2 months
  Percentage of SARS-CoV-2 PCR positive participants (children and educational staff)
Share of participants with SARS-CoV-2 detectable in PCR | 3 months
  Percentage of SARS-CoV-2 PCR positive participants (children and educational staff)
Share of participants with SARS-CoV-2 detectable in PCR | 4 months
  Percentage of SARS-CoV-2 PCR positive participants (children and educational staff)

CONTACTS AND LOCATIONS:
Overall Officials: Nils-Olaf Hübner, Prof. Dr., Principal Investigator — University Medicine Greifswald; Karsten Becker, Prof. Dr., Principal Investigator — University Medicine Greifswald
Locations (1):
- Greifswald University Medicine, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No